CLINICAL TRIAL: NCT01081197
Title: Somatic Disease Among Alcohol Abusers in an Out-day Patients' Clinic. A Neglected Area
Brief Title: Somatic Disease Among Alcohol Abusers in an Out-day Patients' Clinic
Status: Completed | Type: Observational
Sponsor: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: LE_ARP_Somatic_AlcoholAddicts
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: HEART DISEASE; Liver Failure; DEPRESSIVE DISORDER; Alcoholic Neuropathy
Keywords: heart failure; liver; depression; neuropathy
MeSH Terms: conditions — Heart Diseases; Liver Failure; Depressive Disorder; Alcoholic Neuropathy; Heart Failure; Depression | interventions — Psychiatry; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Conventional blood samples including i.e. glycosylated haemoglobin, serum ferritin, serum gamma-GT, B-type natriuretic peptide.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Out-day patients' clinic: Alcohol abusers referred to out-day patients' clinic which consent to participate in the study
  Interventions: Other: Psychiatric and somatic examinations and ,if clinical indicated, treatment
- Control: Control group for the cardiac arm of the study will be matched controls from the Nord-Trøndelag Health Study (HUNT)

INTERVENTIONS:
Other: Psychiatric and somatic examinations and ,if clinical indicated, treatment — Patients referred to the clinic will be given optimal treatment for revealed psychiatric and/or somatic disease including conversational therapy, and if indicated therapeutic interventions with respect to any kind of disease.
  Groups: Out-day patients' clinic

SUMMARY:
Alcohol abuse is associated with a variety of clinical diseases, but studies on prevalence of different somatic diseases among alcohol abusers are lacking. Studies on populations in an out-day patients' clinic are also lacking.

The investigators aim to study somatic health standard in an out-day patients' clinic population of alcohol abusers, with regard to prevalence of different kinds of somatic diseases, and how the interaction of somatic and psychiatric treatment can influence on patients quality of life. Clinical examination including blood samples and echocardiographic examinations in all participants, other additional examinations (as x-ray, CT or MRI if indicated by clinical findings).

DETAILED DESCRIPTION:
Retrospective methods will be used to study former somatic disease, cross-section design to study present somatic disease and prospective design to study quality of life, psychiatric and somatic health after combination of psychiatric and somatic examinations and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol abusers reffered to the out-day patients' clinic at Dep. of Psychiatry, Levanger Hospital, Norway

Exclusion Criteria:

* Not consenting to participate
* Not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alcohol abusers referred to the out-day patients' clinic at Dep. of Psychiatry, Levanger Hospital, Norway
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of different kinds of somatic disease | 3 months after inclusion
  Prevalence of somatic disease at study attendance of any kind, specified for heart disease, gall- and liver disease, neuropathic disease.

SECONDARY OUTCOMES:
Prevalence of former somatic disease | 3 months after inclusion
  Prevalence of former somatic disease investigated by anamnestic examination, search in patient journals and communication with the patients community health service.
Outcome of psychiatric and somatic treatment of alcohol abusers | 1 year after stopped inclusion
  Quality of life and score of somatic and psychiatric health 1 year after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Erling Dalen, MD, Principal Investigator — Helse Nord-Trøndelag HF
Locations (1):
- Levanger Hospital, Dep. of Psychiatry, Levanger, Norway

REFERENCES:
- [Background] Moss M, Parsons PE, Steinberg KP, Hudson LD, Guidot DM, Burnham EL, Eaton S, Cotsonis GA. Chronic alcohol abuse is associated with an increased incidence of acute respiratory distress syndrome and severity of multiple organ dysfunction in patients with septic shock. Crit Care Med. 2003 Mar;31(3):869-77. doi: 10.1097/01.CCM.0000055389.64497.11. PMID 12626999
- [Background] Awtry EH, Philippides GJ. Alcoholic and cocaine-associated cardiomyopathies. Prog Cardiovasc Dis. 2010 Jan-Feb;52(4):289-99. doi: 10.1016/j.pcad.2009.11.004. PMID 20109599
- [Background] Moss M, Burnham EL. Alcohol abuse in the critically ill patient. Lancet. 2006 Dec 23;368(9554):2231-42. doi: 10.1016/S0140-6736(06)69490-7. PMID 17189035
- [Derived] Dalen E, Holmen J, Nordahl HM. Somatic health of patients at an outpatient clinic for substance abuse. Tidsskr Nor Laegeforen. 2015 Jan 27;135(2):127-31. doi: 10.4045/tidsskr.13.0801. eCollection 2015 Jan 27. English, Norwegian. PMID 25625990